CLINICAL TRIAL: NCT04150614
Title: BMT-08: A Comparative Effectiveness Study of the Efficacy and Safety of Transdermal Granisetron to Ondansetron in the Prevention of Nausea and Vomiting in Patients Undergoing Preparative Chemotherapy and Hematopoietic Stem Cell Transplantation
Brief Title: BMT-08: A Comparative Effectiveness Study of Transdermal Granisetron to Ondansetron
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Karen Sweiss, Clinical Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0886
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Nausea With Vomiting Chemotherapy-Induced
Keywords: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to either Arm 1 transdermal granisetron OR Arm 2 intravenous ondansetron
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Active Comparator): ARM 1 -transdermal granisetron plus intravenous dexamethasone
  Interventions: Drug: Granisetron Transdermal Patch; Drug: Intravenous Dexamethasone
- ARM 2 (Active Comparator): ARM 2 -intravenous ondansetron plus intravenous dexamethasone
  Interventions: Drug: Intravenous Dexamethasone; Drug: Ondansetron

INTERVENTIONS:
Drug: Granisetron Transdermal Patch — Antiemetic
  Arms: Arm 1
Drug: Intravenous Dexamethasone — Antiemetic
Drug: Ondansetron — ondansetron
  Arms: ARM 2

SUMMARY:
Patients undergoing either an autologous or allogeneic hematopoietic stem cell transplant (HSCT) and receiving preparative chemotherapy experience a considerable amount of chemotherapy-induced nausea and vomiting (CINV). Current strategies at reducing CINV in this patient population are suboptimal due to lack of efficacy and supportive evidence, potential for increased adverse events, and drug-drug and drug-disease contraindications.

DETAILED DESCRIPTION:
Patients undergoing either an autologous or allogeneic hematopoietic stem cell transplant (HSCT) and receiving preparative chemotherapy experience a considerable amount of chemotherapy-induced nausea and vomiting (CINV). Current strategies at reducing CINV in this patient population are suboptimal due to lack of efficacy and supportive evidence, potential for increased adverse events, and drug-drug and drug-disease contraindications. This study will be an open-label, prospective trial randomizing patients at a 1:1 ratio, to either one of two 5-hydroxytrytamine 3 (5-HT3) antagonists, transdermal granisetron or intravenous (i.v.) ondansetron, in combination with other standard, routinely administered anti-emetic drugs (dexamethasone). Rescue antiemetics will be administered at any time during the study period for vomiting or severe nausea at the request of the patients or as recommended by the attending physicians. For the granisetron treatment arm, patients will be educated and instructed to self-administer a single transdermal granisetron patch one-two days (approximately 24-48 hours) prior to start of the preparative regimen. An additional dose of transdermal granisetron will be administered 7 days after the initial granisetron dose. For the ondansetron treatment arm, patients will receive the standard dose and schedule of intravenous ondansetron that is routinely administered for each respective preparative regimen. Use of rescue medications will be assessed daily during chemotherapy, and for 7 days after the last chemotherapy drug administration (delayed phase). Nausea, vomiting, and treatment-related side effects will be documented and followed during this same time period. A quality of life questionnaire (MDASI-BMT) will be administered at Day + 7 (7 days after day of infusion). All other aspects of patient care (i.e., chemotherapy administration, supportive care, etc.) and laboratory monitoring will adhere to the routine standard of care operating procedures for stem cell transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years at time of enrollment receiving either a preparative regimen and either an autologous or allogeneic stem cell transplant.
* No vomiting ≤ 24 hours prior to registration
* No treatment with an antipsychotic agent such as risperidone, quetiapine, clozapine, phenothiazine or butyrophenone for ≤ 30 days' prior registration or planned during protocol therapy. No patients will be removed from these treatments for study enrollment purposes.
* No chronic phenothiazine administration as an antipsychotic agent (patients may receive prochlorperazine and other phenothiazines as rescue antiemetic therapy). No patients will be removed from these treatments for study enrollment purposes.
* No known hypersensitivity to granisetron

Exclusion Criteria:

* Concurrent use of amifostine
* Known hypersensitivity to granisetron patch or ondansetron
* Patients with a history of long QT syndrome or Torsade de Pointes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To compare between the two study arms the number of patients achieving complete response (no vomiting and no use of rescue medications) during the acute period (0-24 hours post-chemotherapy) for patients receiving preparative chemotherapy and HSCT. | 0 hours to 24 hours post-chemotherapy
  Efficacy of Ondansetron and Dexamethasone versus Transdermal Granisetron and Dexamethasone in preventing chemotherapy induced nausea and vomiting during the acute period (0 - 24 hours post-chemotherapy) for patients receiving preparative chemotherapy and HSCT.

SECONDARY OUTCOMES:
To compare between the two study arms the number of patients achieving complete response (no vomiting and no use of rescue medications) during the delayed period (24-120 hours post-chemotherapy) for patients receiving preparative chemotherapy and HSCT. | 24 hours to 120 hours post-chemotherapy
  Efficacy of Ondansetron and Dexamethasone versus Transdermal Granisetron and Dexamethasone in preventing chemotherapy induced nausea and vomiting during the delayed period (24-120 hours post-chemotherapy) for patients receiving preparative chemotherapy and HSCT.
To compare between the two study arms the number of patients achieving complete response (no vomiting and no use of rescue medications) during the overall period (24-120 hours post-chemotherapy) for patients receiving preparative chemotherapy and HSCT. | 24 hours to 120 hours post-chemotherapy
  Efficacy of Ondansetron and Dexamethasone versus Transdermal Granisetron and Dexamethasone in preventing chemotherapy induced nausea and vomiting during the overall period (24-120 hours post-chemotherapy) for patients receiving preparative chemotherapy and HSCT.
To compare between the two study arms, the use of rescue anti-emetic medications (during and for 7 days after the preparative regimen) for patients receiving preparative chemotherapy and HSCT. | Up to 7 days after the preparative regimen
  Comparing the use of rescue anti-emetic medications between the two arms during and up to 7 days after the preparative regimen
To compare between the two study arms the occurrence of CINV complete protection for patients receiving preparative chemotherapy and HSCT. | Up to 21 - 37 days post-HSCT
  Complete protection is defined as no emetic episode, no use of rescue medications and no nausea, during the acute, delayed, and overall phases
To compare the occurrence of treatment-related adverse events (AE) between patients receiving transdermal Granisetron versus intravenous Ondansetron. | Up to 21 - 37 days post-HSCT
  Treatment-related adverse events (AE) will be evaluated using NCI CTCAE version 5.
To compare quality of life throughout the course of HSCT between patients receiving transdermal Granisetron versus intravenous Ondansetron. | Up to 21-37 days post-HSC
  The M.D. Anderson Symptom Inventory (MDASI) Core Items-Bone Marrow Transplant (BMT) scale will be utilized to measure quality of life at baseline, on the day of stem cell infusion, 7 days after stem cell infusion, and 21-37 days post-stem cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sweiss, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States